CLINICAL TRIAL: NCT03103334
Title: A Single Center Single Dose Open-label Randomized Two Period Crossover Study to Determine the Bioavailability of Two Formulations of Methotrexate 25 mg Administered by Needle Injection and a Pre-filled Needle-free Device in at Least 48 Healthy Volunteers.
Brief Title: A Bioavailability Study of Methotrexate 25 mg Administered by Needle Injection and a Pre Filled Needle-free Device in Healthy Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Crossject (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: L9-E-CJT-CM-131003
Record Dates: First submitted 2017-03-31; First posted 2017-04-06 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Experimental A (Experimental): Zeneo® - Methotrexate thigh to Methotrexate Biodim® thigh
  Interventions: Other: Zeneo® - Methotrexate; Drug: Methotrexate Biodim®
- Experimental B (Experimental): Methotrexate Biodim® thigh to Zeneo® - Methotrexate thigh
  Interventions: Other: Zeneo® - Methotrexate; Drug: Methotrexate Biodim®
- Experimental C (Experimental): Zeneo® - Methotrexate abdomen to Methotrexate Biodim® abdomen
  Interventions: Other: Zeneo® - Methotrexate; Drug: Methotrexate Biodim®
- Experimental D (Experimental): Methotrexate Biodim® abdomen to Zeneo® - Methotrexate abdomen
  Interventions: Other: Zeneo® - Methotrexate; Drug: Methotrexate Biodim®

INTERVENTIONS:
Other: Zeneo® - Methotrexate — 0.625 mL of methotrexate solution 40 mg/ML for subcutaneous injection with a prefilled and needle-free delivery system
Drug: Methotrexate Biodim® — 1 mL of methotrexate solution 25 mg/mL for subcutaneous injection with a conventional needle and syringe injection

SUMMARY:
The objective is to determine whether the test product, Methotrexate 40 mg/mL solution for injection administered subcutaneously by the prefilled and needle-free delivery system Zeneo®, and the reference product, Methotrexate Biodim® 25 mg/mL, solution for injection administered subcutaneously by a conventional syringe with needle are bioequivalent.

DETAILED DESCRIPTION:
ABSTRACT Objective: Zeneo1 is a needle-free injection device. We performed a pharmacokinetic study to investigate the bioequivalence of methotrexate administered subcutaneously using either the needle-free injection device or a conventional needle and syringe.

Research design and methods: This was a single-dose, open-label, laboratory-blind, randomized crossover study performed in adult healthy volunteers. Each participant received two methotrexate injections (each 25mg), one via needle-free injection device and one via conventional injection, with a 21-28 day wash-out interval between dosing. For each participant, the administration site for both injections was either the abdomen or the thigh.

Main outcome measures: The primary pharmacokinetic outcome parameters were AUC(0-t) and Cmax.

Bioequivalence was assessed by standard criteria: whether 90% confidence intervals of geometric mean ratios for the two administration methods were within 80-125%.

Results: Fifty-two individuals completed the study. Bioequivalence criteria were met for AUC(0-t), for the overall analysis (both injection sites: 90% confidence interval: 99.4-103.1%), and for each injection site separately. Bioequivalence was similarly demonstrated with AUC(0-1). Bioequivalence criteria for Cmax were fulfilled for abdominal administration but not for the overall analysis. Injection via the needle- free injection device was well tolerated.

Limitations: Limitations include conducting the study in healthy volunteers and the relatively small subject number (albeit satisfactory for bioequivalence).

Conclusions: This study shows that methotrexate injection via needle-free injection device is bioequivalent to a conventional needle and syringe in relation to AUC(0-t) and AUC(0-1). Studies of needle-free injection device use in patients requiring methotrexate therapy are planned.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* BMI between 18.5 and 30 kg/m2
* Body mass > 60 kg
* Non-tobacco user
* Written consent given for participation in the study

Exclusion Criteria:

* Evidence of clinically relevant oral, cardiovascular, hematologic, gastrointestinal, hepatic, renal, endocrine, pulmonary, neurologic, psychiatric or skin disorder
* Heavy alcohol consumption and regular exposure to drug of abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2014-06; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax). | serial pharmacokinetic plasma concentrations were drawn prior pre-dose and post-dose at 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16 and 24 hours
Area under the plasma concentration versus time curve (AUC) time zero to time of the last quantifiable concentration (AUC(0-t)). | serial pharmacokinetic plasma concentrations were drawn prior pre-dose and post-dose at 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16 and 24 hours

IPD SHARING:
Plan to Share IPD: No